CLINICAL TRIAL: NCT05251857
Title: Animation Education Program Applied to Laparoscopic Sleeve Gastrectomy Patients Effect on Patient Care Results: A Randomized Controlled Trial
Brief Title: Animation Education Program Applied to Laparoscopic Sleeve Gastrectomy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ayşegül Yayla, Asistant Professors, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AEP16
Record Dates: First submitted 2021-12-29; First posted 2022-02-23 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Surgery; Educational Problems

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Animation Education Program Applied to Laparoscopic Sleeve Gastrectomy Patients (Experimental): The intervention group is the group in which the investigors applied animation education program Intervention: Behavioral: Animation Education Program
  Interventions: Behavioral: Animation Education Program Applied to Laparoscopic Sleeve Gastrectomy Patients
- Standard Clinical Care Applied to Laparoscopic Sleeve Gastrectomy Patients (No Intervention): The control group is the group that receives standard clinical care

INTERVENTIONS:
Behavioral: Animation Education Program Applied to Laparoscopic Sleeve Gastrectomy Patients — Behavioral: Animation Education Program The investigators will apply Animation Education Program.
  Arms: Animation Education Program Applied to Laparoscopic Sleeve Gastrectomy Patients

SUMMARY:
Objectives This study investigated the effect of animation education developed for respiratory rehabilitation among sleeve gastrectomy patients on patient care results.

Design This is a randomized controlled study. Method A total of 66 patients who were going to have sleeve gastrectomy were randomly divided into two groups each including 33 participants. The intervention group was provided with animation education. The control group received routine face-to-face education. Postoperative risk of respiratory complications, presence of dyspnea, nausea, and vomiting, frequency of postoperative respiratory exercises, and satisfaction with postoperative respiratory education were examined. Patients' pain and sleep quality were examined one day before the surgery and on the postoperative first and fifth days.

ELIGIBILITY:
Inclusion Criteria:

The patients,

who are in clinical treatment for sleeve gastrectomy; who are 18 years of age or older, mentally healthy; who can speak and understand Turkish; who owns and can use smartphones; who do not have chronic diseases related to the respiratory system (lung diseases, etc.); who are volunteers, will be included in the study.

Exclusion Criteria:

The Patients

who are a lung infection in the last month who are neurological disease who are major psychiatric diagnosis who are vision and hearing problems who are intolerable dyspnea who do not agree to participate in the study, will be excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | until the treatment is completed,an average of 5 days
  Pain levels Visual Analog Scale (VAS): The VAS was used to evaluate the severity of pain in patients. VAS is a 10 cm ruler that shows no pain on one edge and unbearable pain on the other edge. Therefore, patients are asked to evaluate their pain between 0 "no pain" and 10 "unbearable pain." They show the severity of their pain using a sign on that ruler. The point indicated by the patient is recorded from the starting point of 0. VAS is an understandable and easily applicable scale to evaluate the pain levels of patients
Richard Campbell Sleep Questionnaire (RCSQ) | until the treatment is completed,an average of 5 days
  Sleep quality Richard Campbell Sleep Questionnaire (RCSQ) The scale was developed by Richards in 1987. Its Turkish validity and reliability study was conducted by Özlü and Özer in 2015. RCSQ evaluates the depth of night sleep, time to fall asleep, frequency of awakening, time awake when awakened, sleep quality, and the noise level in the environment. The scale consists of 6 questions. Each item is scored between 0 and 100 using the VAS. A score of 0-25 points obtained from the scale indicates very bad sleep and 76-100 indicates very good sleep.

SECONDARY OUTCOMES:
Respiratory complications question form | until the treatment is completed,an average of 5 days
  respiratory complications

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yayla A, Menevse S. Animation Education Program Applied to Laparoscopic Sleeve Gastrectomy Patients Effect on Patient Care Results: A Randomized Controlled Trial. Clin Nurs Res. 2023 Jan;32(1):126-137. doi: 10.1177/10547738221112754. Epub 2022 Aug 23. PMID 36000187